CLINICAL TRIAL: NCT01051882
Title: A Phase I/II, Open Label Study to Evaluate Safety, Tolerability and Therapeutic Effects of Transplantation of Autologous Cultured Mesenchymal Bone Marrow Stromal Cells Secreting Neurotrophic Factors (MSC-NTF), in ALS Patients.
Brief Title: Autologous Cultured Mesenchymal Bone Marrow Stromal Cells Secreting Neurotrophic Factors (MSC-NTF), in ALS Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-NTF-001-HMO-CTIL
Record Dates: First submitted 2010-01-17; First posted 2010-01-20 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2012-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Mesenchymal Stromal Cells (MSC); Amyotrophic Lateral Sclerosis (ALS); Neuroprotection; Neurodegeneration; Stem cells; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nerve Degeneration

ARMS (2):
- MSC-NTF cells IM (Experimental): Intramuscular administration in early stage patients
  Interventions: Biological: MSC-NTF cells transplantation (IM)
- MSC-NTF cells IT (Experimental): Intrathecal administration in progressive stage patients
  Interventions: Biological: MSC-NTF cells transplantation (IT)

INTERVENTIONS:
Biological: MSC-NTF cells transplantation (IM) — In early ALS subjects: Autologous MSC-NTF cells will be transplanted under mild anesthesia, intramuscularly into patients' clinically unaffected (or only mildly affected) upper arm biceps and triceps muscles according to a pre-designed grid. Intramuscular injections will be by a 26 gauge needle to a 1.5cm depth (ensuring that injection is into muscle and not adipose tissue). The patients will be injected at 24 sites with a total of 24 million cells
  Arms: MSC-NTF cells IM
Biological: MSC-NTF cells transplantation (IT) — In progressive ALS subjects: Autologous MSC-NTF cells will be transplanted under mild anesthesia intrathecally(via a standard lumbar puncture)with a total of 60 million cells.
  Arms: MSC-NTF cells IT

SUMMARY:
The study will evaluate the safety, tolerability and therapeutic effects (preliminary efficacy) of injection of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF), as a possible treatment for patients with Amyotrophic Lateral Sclerosis (ALS) at the early and progressive disease stages.

DETAILED DESCRIPTION:
This study is a single center trial to be conducted at the Department of Neurology & Laboratory of Neuroimmunology, at the Hadassah Hebrew University Medical Center, Jerusalem in Israel. All patients enrolled will have a documented history of ALS disease prior to study enrolment. Patients diagnosed as early stage ALS disease with duration of less than 6 months and patients diagnosed with progressive stage ALS disease with duration of 6-12 months. Overall, 24 patients will be recruited and allocated based on their ALS disease severity to 2 treatment groups: Group A - 12 patients of early ALS disease stage and Group B - 12 patients of progressive ALS disease.

Eligible patients will be enrolled into the study and will be observed for every 2 weeks during a "run in period" of 3 months for determination of the progression rate of the disease. During the "run in period" after about 6 weeks following enrollment, patients of both study groups will undergo a Bone Marrow Aspiration procedure and MSC-NTF cells will be produced from the bone marrow aspirate based on Brainstorm Cell Therapeutics Ltd proprietary method. On the last "run in period" visit, patients of both study groups will undergo the treatment and MSC-NTF will be transplanted by IM or IT injection to the early and progressive ALS patients respectively.

After the MSC-NTF transplantation patients will be observed on a monthly basis for a post treatment follow up period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. El Escorial criteria for definite or probable ALS
2. Either men or non pregnant women between 20-75 years of age.
3. Patient is mentally intact and psychologically stable
4. For early stage ALS- Patients will be with ALS-FRS-R scale of at least 30 and disease duration of less than 2 years.Or, for progressive stage ALS- Patients will be with an ALS-FRS-R scale of 15-30 and disease duration of less than 2 years
5. For early stage ALS- Patient has sufficiently bulky muscles. Or, for progressive stage ALS- Patient with at least 60% FVC
6. Participant understands the nature of the procedure and provides written informed consent prior to any study procedure.

Exclusion Criteria:

1. Positive test for HBV, HCV, HIV and Mycoplasma.
2. High protein in the CSF.
3. Lymphocytosis in the CSF.
4. Positive for anti-GM1 antibodies.
5. Patient has significant conduction blocks or slow nerve conduction velocities (a reduction of more than 30%) confirmed by nerve conduction velocity - EMG studies.
6. The patient is a respiratory dependent.
7. Renal failure, impaired hepatic function
8. Patients suffering from significant cardiac disease, malignant diseases or any other disease that may risk the patient or interfere with the ability to interpret the results
9. Active infections.
10. Participation in another clinical trial within 1 month prior to start of this study.
11. Subject unwilling or unable to comply with the requirements of the protocol.
12. Patient has not been treated previously with any cellular therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety evaluation and tolerability of a single treatment administration of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF) | 6 months
  Safety evaluation and tolerability of a single treatment administration of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF) by multiple intramuscular injections (IM) at 24 separate sites on the biceps and triceps muscles to patients with ALS at the early disease stage
Safety evaluation and tolerability of single intrathecal injection (IT) into the cerebrospinal fluid (CSF) of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF) | 6 months
  Safety evaluation and tolerability of single intrathecal injection (IT) into the cerebrospinal fluid (CSF) of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF),to patients with ALS at the progressive disease stage.

SECONDARY OUTCOMES:
Changes in the progression rate of the disease as evidenced by changes in the ALS functional rating scale (ALS-FRS) | 6 months
Changes in muscle strength grading (MVIC) by muscle chart | 6 months
Changes in forced vital capacity (FVC %) (In the progressive disease stage group only). | 6 months
Changes in muscle bulk estimated by MRI of the upper and lower extremities | 6 months
Changes in upper and lower extremities circumference (cm) | 6 months
Changes in EMG parameters | 6 months
Need and time to tracheotomy or permanent assisted ventilation | 6 months
Overall survival, calculating time to death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karussis, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Petrou P, Gothelf Y, Argov Z, Gotkine M, Levy YS, Kassis I, Vaknin-Dembinsky A, Ben-Hur T, Offen D, Abramsky O, Melamed E, Karussis D. Safety and Clinical Effects of Mesenchymal Stem Cells Secreting Neurotrophic Factor Transplantation in Patients With Amyotrophic Lateral Sclerosis: Results of Phase 1/2 and 2a Clinical Trials. JAMA Neurol. 2016 Mar;73(3):337-44. doi: 10.1001/jamaneurol.2015.4321. PMID 26751635